CLINICAL TRIAL: NCT05432466
Title: A Phase 3 Randomized, Double-Blind, Decentralized Clinical Trial to Compare the Efficacy of Celiprolol to Placebo in the Treatment of Patients With COL3A1-Positive Vascular Ehlers-Danlos Syndrome
Brief Title: Clinical Trial to Compare the Efficacy of Celiprolol to Placebo in Patients With Vascular Ehlers-Danlos Syndrome
Acronym: DiSCOVER
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Acer Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACER-002-301
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Vascular Ehlers-Danlos Syndrome
MeSH Terms: conditions — Ehlers-Danlos Syndrome, Type IV | interventions — Celiprolol; BID protein, human

STUDY DESIGN:
Intervention Model Description: This is a prospective, Phase 3, randomized, double-blind, placebo-controlled efficacy study to evaluate celiprolol in patients genetically confirmed as COL3A1-positive vEDS using a decentralized clinical trial design.
  The double-blind portion of this study is intended to end at Month 40 assuming that at least 46 vEDS-related clinical events have occurred. If the number of vEDS-related events is fewer than 46 at Month 40, the study will continue until the required number of events have occurred prior to ending the double-blind portion of the study.
  Following the double-blind treatment period or occurrence of a vEDS-related clinical event, patients have the option to participate in an OLE period.
  A total of approximately 150 patients who meet all the inclusion and none of the exclusion criteria will be enrolled and randomized 2:1 to receive either celiprolol or placebo, respectively.
  An approximately 40-month treatment period followed by an optional open-label extension study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient, the Investigator, and other members of the staff involved with the study will remain blinded to the two study treatments (celiprolol and placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ACER-002 (celiprolol) 200 mg BID (Experimental): ACER-002 200 mg twice daily (BID) (after titration):
  200 mg morning and 200 mg evening: 400 mg total daily dose
  Titration:
  Day 1 to Month 1 - 100 mg once daily (QD) evening: 100 mg total daily dose Month 2 to Month 3 - 100 mg morning and 100 mg evening: 200 mg total daily dose Month 3 to Month 4 - 100 mg morning and 200 mg evening: 300 mg total daily dose Month 4 to End of Treatment Period (BID) - 200 mg morning and 200 mg evening: 400 mg total daily dose
  Interventions: Drug: ACER-002 (celiprolol) 200 mg BID
- Placebo BID (Experimental): Placebo twice daily (BID) Placebo given orally to mimic ACER-002 (celiprolol) administration
  Interventions: Drug: Placebo BID

INTERVENTIONS:
Drug: ACER-002 (celiprolol) 200 mg BID — ACER-002 (celiprolol) 200 mg BID
  Other Names: ACER-002; celiprolol
  Arms: ACER-002 (celiprolol) 200 mg BID
Drug: Placebo BID — placebo for ACER-002
  Other Names: placebo
  Arms: Placebo BID

SUMMARY:
This is a prospective, Phase 3, randomized, double-blind, placebo-controlled efficacy study to evaluate celiprolol in patients genetically confirmed as COL3A1-positive vEDS using a decentralized clinical trial design.

DETAILED DESCRIPTION:
This is a prospective, Phase 3, randomized, double-blind, placebo-controlled efficacy study to evaluate celiprolol in patients genetically confirmed as COL3A1-positive vEDS using a decentralized clinical trial design.

The double-blind portion of this study is intended to end if statistical significance is reached at the interim analysis (accrual of 28 vEDS-related events requiring medical attention; estimated to take 24 months) or after accrual of 46 vEDS related clinical events requiring medical attention (estimated to take 40 months).

A total of approximately 150 patients who meet all the inclusion and none of the exclusion criteria will be enrolled and randomized 2:1 to receive either celiprolol or placebo, respectively.

Following the double-blind treatment period or occurrence of vEDS-related clinical event, patients have the option to participate in an open label extension period.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to obtain magnetic resonance angiogram (MRA) image at local imaging facility.
2. A genetic test confirming the presence of a pathogenic COL3A1 variant (classified as likely pathogenic or pathogenic according to ACMG/AMP Guidelines.
3. Patients must be ≥ 15 years of age at the time of randomization.
4. Able and willing to discontinue use of β-blockers prior to randomization.

Exclusion Criteria:

1. Lack of a COL3A1-positive test at screening (e.g., COL3A1 benign, likely benign, variant of unknown significance [VUS] or no variant) or presence of a COL3A1 variant but demonstration of a COL3A1 variant reported to be a haploinsufficiency variant.
2. Arterial rupture or dissection, uterine rupture, and/or intestinal rupture within 6 months prior to Screening.
3. Patients unable to discontinue β-blocker treatment prior to randomization.
4. Unable or unwilling to complete the study procedures.
5. Breastfeeding, pregnancy, or planned pregnancy during the trial.
6. Any medical condition that in the opinion of the Investigator may pose a safety risk to the patient in this study, which may confound efficacy or safety assessment, or may interfere with study participation.
7. Use of any prohibited medications

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of a vEDS-related clinical event requiring medical attention: Fatal/nonfatal cardiac or arterial events [including dissection or rupture], uterine rupture, intestinal rupture, and/or unexplained sudden death | Over the double-blind period (estimated to be 40 months)

SECONDARY OUTCOMES:
Number and proportion of patients reporting a vEDS related clinical event requiring medical attention: Fatal/nonfatal cardiac or arterial events [including dissection or rupture], uterine rupture, intestinal rupture, and/or unexplained sudden death | Over the double-blind period (estimated to be 40 months)
Number and percentage of patients with adverse events | Over the double-blind period (estimated to be 40 months)
  An Adverse Event (AE) is defined as any untoward medical occurrence associated with the use of the investigational product in humans, whether or not considered related to investigational product. An AE can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with any use of the investigational product, without any judgment about causality and irrespective of route of administration, formulation, or dose, including an overdose.
Number and percentage of Serious Adverse Events (SAE) | Over the double-blind period (estimated to be 40 months)
  An AE is considered "serious" if, in the view of either the investigator or Acer, it results in any of the following outcomes: Death, Is immediately life threatening; Requires in-patient hospitalization or prolongation of existing hospitalization; Results in persistent or significant disability or incapacity; Results in a congenital abnormality or birth defect; Is an important medical event that may jeopardize the subject or may require medical intervention to prevent one of the outcomes listed above.
Number and percentage of patient deaths | Over the double-blind period (estimated to be 40 months)
Number and percentage of patient discontinuations | Over the double-blind period (estimated to be 40 months)
  Discontinuation or withdrawal from the study

CONTACTS AND LOCATIONS:
Locations (1):
- Science 37, Culver City, California, United States

IPD SHARING:
Plan to Share IPD: No